CLINICAL TRIAL: NCT07088978
Title: Adaptation of the Patient Reported Outcomes for Fighting Financial Toxicity of Cancer (PROFFIT) Instrument Into Turkish: A Validity and Reliability Study
Brief Title: Adaptation of the PROFFIT Instrument Into Turkish: A Validity and Reliability Study
Status: Not yet recruiting | Type: Observational
Sponsor: Akdeniz University (Other)
Collaborators: Giresun Training and Research Hospital (Unknown); St. Mary's University, Twickenham (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network)
Responsible Party: Principal Investigator, Zeynep KARAKUŞ, Research Assistant, PhD, Akdeniz University
Other Study IDs: Akdeniz_University
Record Dates: First submitted 2025-06-02; First posted 2025-07-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the Turkish validity and reliability of the Patient Reported Outcomes for Fighting Financial Toxicity of Cancer (PROFFIT) developed in Italy.

DETAILED DESCRIPTION:
The scale validity of the study will be evaluated through language and content validity, construct validity, criterion validity, and known-group validity methods; while the scale reliability will be assessed by calculating the Cronbach's alpha and McDonald's omega reliability coefficients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with solid cancer or hematologic malignancy, either histologically or cytologically, and aware of their diagnosis,
* Those who have received cancer treatment (chemotherapy, targeted therapy, immunotherapy, hormonal therapy, radiotherapy, or a combination of these treatments) within the last three months,
* Individuals over the age of 18,
* Those without a diagnosed psychiatric illness (such as depression, panic attacks, schizophrenia, etc.),
* Individuals without auditory or cognitive impairments,
* Turkish-speaking and literate volunteers.

Exclusion Criteria:

* Individuals who fill out the data collection forms incompletely or wish to withdraw from the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Turkish-speaking and literate volunteers over the age of 18 diagnosed with solid cancer or hematologic malignancy who have received cancer treatment (chemotherapy, targeted therapy, immunotherapy, hormonal therapy, radiotherapy, or a combination of these treatments) within the last three months.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Validity Assessment-Language and Content Validity | Through study completion, an average of 12 months
  Language and Content Validity: To assess the relevance and appropriateness of the translated items, a panel of at least six experts in oncology, psychology, and instrument development will evaluate each item.
Validity Assessment-Content Validity Index (CVI) | Through study completion, an average of 12 months
  Content Validity Index (CVI) will be calculated based on expert ratings to determine the proportion of items deemed relevant.
Validity Assessment-Content Validity Ratio (CVR) | Through study completion, an average of 12 months
  Content Validity Ratio (CVR) will be used to assess whether each item is essential for measuring the construct.
Validity Assessment-Construct Validity | Through study completion, an average of 12 months
  Confirmatory Factor Analysis (CFA) will be performed to verify whether the factor structure of the Turkish version aligns with that of the original instrument.
  Model fit indices such as χ²/df, RMSEA, CFI, TLI, and SRMR will be used to evaluate the adequacy of the factor structure.
Validity Assessment- Criterion Validity | Through study completion, an average of 12 months
  The Turkish PROFFIT scores will be correlated with other established patient-reported outcome measures, specifically the COST (v2) and EORTC QLQ-C30 instruments, to assess convergent validity.
  Pearson or Spearman correlation coefficients will be used to determine the strength of associations between PROFFIT and these validated measures.
Validity Assessment- Known-Group Validity | Through study completion, an average of 12 months
  To assess whether the instrument can differentiate between groups with known differences in financial toxicity, mean scores of the total and subscales will be compared across predefined demographic and clinical groups.
  Independent samples t-tests and ANOVA will be performed to compare group differences.
Reliability Assessment | Through study completion, an average of 12 months
  Internal Consistency: The reliability of the Turkish PROFFIT instrument will be evaluated using:
  Cronbach's alpha (α) to assess the overall internal consistency of the scale. McDonald's omega (ω) as an alternative measure that provides a more robust estimation of reliability in multidimensional scales.

IPD SHARING:
Plan to Share IPD: Undecided